CLINICAL TRIAL: NCT00674375
Title: Can Risk Score Alerts Improve Office Care for Chest Pain?
Brief Title: Risk Score Alerts for Chest Pain Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard Vanguard Medical Associates (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Thomas Dean Sequist, Principal Investigator, Harvard Vanguard Medical Associates
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R18HS017075-01 (AHRQ)
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Chest Pain; Acute Myocardial Infarction
Keywords: Chest Pain; Acute Myocardial Infarction; Patient Safety; Misdiagnosis
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Primary care clinicians (physicians, nurse practitioners, and physician assistants) randomized to the intervention arm will receive electronic alerts within the electronic medical record system during office visits with patients complaining of chest pain.
  Interventions: Other: Electronic risk alerts
- 2 (No Intervention): Primary care clinicians randomized to the 'no intervention' arm will evaluate and treat patients complaining of chest pain without the aid of electronic risk alerts.

INTERVENTIONS:
Other: Electronic risk alerts — Electronic risk alerts within the electronic medical record system will automatically calculate a patient's Framingham Risk Score during office visits for chest pain. These alerts will recommend electrocardiogram performance and aspirin therapy for patients with Framingham Risk Score at least 10%, and will recommend against exercise stress testing for patients with a Framingham Risk Score less than 10%.
  Arms: 1

SUMMARY:
The evaluation of chest pain in the primary care office is a challenging problem, with many patients suffering from missed diagnoses of acute myocardial infarction and many other low risk patients receiving unnecessary evaluations. This project will provide primary care physicians evaluating patients complaining of chest pain with computerized alerts that differentiate high-risk patients from low risk patients, and provide individualized evaluation and treatment recommendations.

DETAILED DESCRIPTION:
The evaluation of ambulatory patients with chest pain is a challenging and serious problem, accounting for a significant proportion of all outpatient visits. High risk patients may go undetected, resulting in missed diagnoses of acute myocardial ischemia, while low risk patients may be subject to unnecessary evaluations. To substantially improve the evaluation and treatment of outpatients with acute chest pain syndromes, new strategies need to be developed in the primary care setting to risk stratify symptomatic patients and direct appropriate care. Our prior work demonstrates that an elevated Framingham Risk Score (at least 10%) reliably identifies patients with chest pain in the primary care setting who are at high risk for acute myocardial infarction.

This study will implement and evaluate electronic risk alerts to risk stratify outpatients with chest pain and present this information to primary care clinicians within the context of an electronic health record. The intervention will take place within Harvard Vanguard Medical Associates, a multispecialty integrated group practice with 140 primary care physicians caring for approximately 300,000 patients at 14 centers in eastern Massachusetts. With a randomized, controlled study design, the study has three specific aims:

* To identify predictors of risk-appropriate evaluation and treatment of patients presenting to primary care offices with acute chest pain, including race and sex.
* To determine whether rates of appropriate evaluation and treatment of patients with acute chest pain can be improved through the use of point-of-care electronic risk alerts that provide individual patient cardiac risk profiles and tailored evaluation and treatment recommendations to primary care clinicians.
* To perform a cost analysis for the provision of electronic decision support for patients with acute chest pain.

This study has important implications for determining how the treatment of outpatients with chest pain syndromes can be optimized through the innovative use of electronic decision support, while documenting the cost implications of such a strategy. This work will also provide a model for how ambulatory practices across the country can use electronic health records to present real-time patient risk information to clinicians with the goal of improving patient safety and quality, which has important implications for both acute and chronic care.

ELIGIBILITY:
Inclusion Criteria:

* Adults 30 years and older presenting to one of 14 ambulatory health centers and their evaluating primary care clinician will be eligible for this study.

Exclusion Criteria:

* Prior history of coronary heart disease
* Age <30 years
* Presentation for an annual physical examination
* Prior hospital admission or emergency department visit for evaluation of chest pain within 30 days of their presentation to primary care clinician

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Performance of electrocardiogram for patients with Framingham Risk Score greater than or equal to 10%. | During office visit
Administration of aspirin therapy for patients with Framingham Risk Score greater than or equal to 10% | During office visit
Performance of exercise stress testing for patients with Framingham Risk Score less than 10% | Within 2 months of office visit

SECONDARY OUTCOMES:
EKG and aspirin therapy for patients with Framingham Risk Score at least 10% among intervention and control clinicians according to clinician risk tolerance. Hypothesis: Intervention effect will be greatest among clinicians with a high risk tolerance. | During office visit
Exercise stress testing for patients with Framingham Risk Score less than 10% among intervention and control clinicians according to clinician risk tolerance. Hypothesis: Intervention effect will be greatest among clinicians with lowest risk tolerance. | Within 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Sequist, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Newton, Massachusetts

REFERENCES:
- [Background] Sequist TD, Marshall R, Lampert S, Buechler EJ, Lee TH. Missed opportunities in the primary care management of early acute ischemic heart disease. Arch Intern Med. 2006 Nov 13;166(20):2237-43. doi: 10.1001/archinte.166.20.2237. PMID 17101942
- [Derived] Sequist TD, Morong SM, Marston A, Keohane CA, Cook EF, Orav EJ, Lee TH. Electronic risk alerts to improve primary care management of chest pain: a randomized, controlled trial. J Gen Intern Med. 2012 Apr;27(4):438-44. doi: 10.1007/s11606-011-1911-6. Epub 2011 Oct 13. PMID 21993999
- See also: Harvard Vanguard Medical Associates — http://www.harvardvanguard.org